CLINICAL TRIAL: NCT04947306
Title: A Comparison of Accelerometric Monitoring by TOF Watch® SX and Electromyographic Monitoring by Tetragraph® for Recovery From Neuromuscular Blockade
Brief Title: A Comparison Between TOF Watch® SX and Tetragraph®
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: INT58/20
Record Dates: First submitted 2021-06-15; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Neuromuscular Blockade; Neuromuscular Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects: Adult patients >18 years of age, who are scheduled to undergo any elective procedure under general anesthesia at our Institution in which the administration of rocuronium for neuromuscular blockade is anticipated.
  All participants will be monitored with both TOF Watch and Tetragraph neuromuscular monitors.
  Interventions: Device: Tetragraph® (Senzime, Uppsala, Sweden); Device: TOF Watch® SX (Organon Teknika B.V., Boxtel, Holland)

INTERVENTIONS:
Device: Tetragraph® (Senzime, Uppsala, Sweden) — The Tetragraph® is a recently marketed electromyographic neuromuscular monitor that uses a disposable electrode array (TetraSens) that combines stimulating and recording electrodes
  Other Names: Electromyographic neuromuscular monitor
Device: TOF Watch® SX (Organon Teknika B.V., Boxtel, Holland) — The TOF Watch® SX is a common used neuromuscular monitor
  Other Names: Acceleromyographic neuromuscular monitor

SUMMARY:
This observational study was designed to assess the agreement between the recently marketed electromyographic neuromuscular blockade monitor Tetragraph® (Senzime, Uppsala, Sweden) and the TOF Watch® SX (Organon Teknika B.V., Boxtel, Holland), an accelerometric neuromuscular blockade monitor frequently used in clinical practice

DETAILED DESCRIPTION:
Before the induction of general anesthesia both monitors will be placed in the same arm. After induction of general anesthesia and before neuromuscular blocking agent administration both devices will be consecutively calibrated and a baseline measurement will be obtained. During the surgical procedure the investigators will monitor neuromuscular function with one of the two devices. Then the investigators will switch the device used as a guide between subsequent patients. The protocol will start as soon as the leading device will register a train-of-four ratio (TOFr) ≥ 0.2. During the protocol a comparison between the two devices will be conducted as soon as the device used as a guide will display a TOFr ≥ 0.2, 0.3, 0.4, 0.5, 0.6, 0.7, 0.8, 0.9, 1. For each of the TOFr reported, we will deliver two subsequent TOF stimulations with the guiding device followed by two TOF stimulations with the other monitor. Both the stimulations delivered by each device and the two consecutive stimulations delivered by different monitors will be conducted 20 sec from one another. Stimulations with the same device will be used to assess intraobserver variability for each methodology, while the second and the third measurements (consecutive stimulations with different devices) will be used to assess agreement between them. The protocol will end when the leading device will show a TOFr ≥ 1.0, or if, at the end of the surgical procedure, acceleromyographic TOFr will be > 0.9.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Rocuronium bromide use is anticipated for neuromuscular blockade during surgical procedure
* Upper arms will be freely available during the surgical procedure

Exclusion Criteria:

* Known neuromuscular disease
* Known allergy to Rocuronium bromide
* end-stage liver disease
* chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients >18 years of age, who are scheduled to undergo any elective procedure under general anesthesia at our Institution in which the administration of rocuronium for neuromuscular blockade is anticipated.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Agreement between TOF Watch® SX and Tetragraph® train-of-four ratios | Recovery from neuromuscular blockade at the end of the surgical procedure
  Bias and Limits of Agreement between the two methodologies using Bland-Altman analysis

SECONDARY OUTCOMES:
Agreement between normalized TOF Watch® SX and Tetragraph® train-of-four ratios | Recovery from neuromuscular blockade at the end of the surgical procedure
  Normalized TOF Watch® SX train of four ratios will be calculated as the ratio between actual train-of-four ratio and baseline. Bias and Limits of Agreement will be derived using Bland-Altman analysis
Agreement between TOF Watch® SX and Tetragraph® train-of-four ratios for TOF ratios < 0.8 | Recovery from neuromuscular blockade at the end of the surgical procedure
  Normalized TOF Watch® SX train of four ratios will be calculated as the ratio between actual train-of-four ratio and baseline. Bias and Limits of Agreement will be derived using Bland-Altman analysis
Agreement between TOF Watch® SX and Tetragraph® train-of-four ratios for TOF ratios ≥ 0.8 | Recovery from neuromuscular blockade at the end of the surgical procedure
  Normalized TOF Watch® SX train of four ratios will be calculated as the ratio between actual train-of-four ratio and baseline. Bias and Limits of Agreement will be derived using Bland-Altman analysis
Absolute and relative intraobserver variability for TOF Watch® SX and Tetragraph® | Recovery from neuromuscular blockade at the end of the surgical procedure
  Absolute intraobserver variability will be calculated as the absolute difference between pairs of consecutive measurements by the same device. Relative intraobserver variability will be calculated as the ratio between the absolute difference and mean of the measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No